CLINICAL TRIAL: NCT05826301
Title: Percutaneous Neuromodulation in Tibial Nerve vs. Electrolysis in Plantar Fasciitis Subjects
Brief Title: Neuromodulation vs. Electrolysis in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA-11/8/HMC/DADCI
Record Dates: First submitted 2023-02-21; First posted 2023-04-24 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-04

CONDITIONS: Plantar Fascitis
Keywords: pain; plantar fasciitis; ultrasound imaging; quality of life
MeSH Terms: conditions — Pain; Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous neuromodulation in tibial nerve (Experimental): Specifically, the procedure consisted in the application of a square wave biphasic electrical current, with 2-4 Hz frequency, 450 μs pulse during 25 minutes with a needle (0.30mm x 40 mm) inserted proximal to the surface on the tibial nerve.
  2 times per week
  Interventions: Other: Percutaneous neuromodulation in tibial nerve
- Percutaneous electrolysis (Active Comparator): The procedure consist on placed a needle (0.30mm x 40 mm) on the most hyperalgesic plantar fascia location with a galvanic current of 3mA, 3 times during 3 seconds.
  1 time per week
  Interventions: Other: Percutaneous electrolysis

INTERVENTIONS:
Other: Percutaneous neuromodulation in tibial nerve — The procedure consisted in the application of a square wave biphasic electrical current, with 2-4 Hz frequency, 450 μs pulse during 25 minutes with a needle (0.30mm x 40 mm) inserted proximal to the surface on the tibial nerve.
  Arms: Percutaneous neuromodulation in tibial nerve
Other: Percutaneous electrolysis — The procedure consist on placed a needle (0.30mm x 40 mm) on the most hyperalgesic plantar fascia location with a galvanic current of 3mA, 3 times during 3 seconds.
  1 time per weeK
  Arms: Percutaneous electrolysis

SUMMARY:
The aim of the present study will be the implementation of two protocols in plantar fasciitis individuals: a) percutaneous neuromodulation, b) percutaneous electrolysis in plantar fascia. Authors hypothesized that percutaneous neuromodulation may have benefits in: pain, quality of life, muscular structure.

ELIGIBILITY:
Inclusion Criteria:

* Patiens with plantar fasciitis

Exclusion Criteria:

* Lower limb disturbances
* Sistemic diseases
* Not involved in other drug or manual therapy interventions
* Infections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Pre intervention
  visual analoge scale (VAS)
Pain intensity | immediately post intervention
  visual analogue scale (VAS)
Pain intensity | at 4 weeks
  visual analogue scale (VAS)

SECONDARY OUTCOMES:
quality of life perception | Pre intervention
  SF-36 questionnaire
quality of life perception | immediately post intervention
  SF-36 questionnaire
quality of life perception | at 4 weeks
  SF-36 questionnaire
Ultrasonography of extrinsic foot muscles | Pre intervention
  Ultrasound imaging of the thickness and cross-sectional area of the tibiais
Ultrasonography of extrinsic foot muscles | immediately post intervention
  Ultrasound imaging of the thickness and cross-sectional area of the tibiais
Ultrasonography of extrinsic foot muscles | at 4 weeks
  Ultrasound imaging of the thickness and cross-sectional area of the tibiais

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - UEM, Madrid
  - Universidad Europea, Madrid

REFERENCES:
- [Background] De-la-Cruz-Torres B, Abuin-Porras V, Navarro-Flores E, Calvo-Lobo C, Romero-Morales C. Ultrasound-Guided Percutaneous Neuromodulation in Patients with Chronic Lateral Epicondylalgia: A Pilot Randomized Clinical Trial. Int J Environ Res Public Health. 2021 May 3;18(9):4877. doi: 10.3390/ijerph18094877. PMID 34063673
- [Background] Ilfeld BM, Gelfand H, Dhanjal S, Hackworth R, Plunkett A, Turan A, Vijjeswarapu AM, Cohen SP, Eisenach JC, Griffith S, Hanling S, Mascha EJ, Sessler DI. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: A Pragmatic Effectiveness Trial of a Nonpharmacologic Alternative for the Treatment of Postoperative Pain. Pain Med. 2020 Dec 12;21(Suppl 2):S53-S61. doi: 10.1093/pm/pnaa332. PMID 33313729
- [Background] Ilfeld BM, Said ET, Finneran JJ 4th, Sztain JF, Abramson WB, Gabriel RA, Khatibi B, Swisher MW, Jaeger P, Covey DC, Robertson CM. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Femoral Nerve for Postoperative Analgesia Following Ambulatory Anterior Cruciate Ligament Reconstruction: A Proof of Concept Study. Neuromodulation. 2019 Jul;22(5):621-629. doi: 10.1111/ner.12851. Epub 2018 Aug 30. PMID 30160335
- [Background] Ilfeld BM, Gilmore CA, Grant SA, Bolognesi MP, Del Gaizo DJ, Wongsarnpigoon A, Boggs JW. Ultrasound-guided percutaneous peripheral nerve stimulation for analgesia following total knee arthroplasty: a prospective feasibility study. J Orthop Surg Res. 2017 Jan 13;12(1):4. doi: 10.1186/s13018-016-0506-7. PMID 28086940
- [Background] San-Emeterio-Iglesias R, Minaya-Munoz F, Romero-Morales C, De-la-Cruz-Torres B. Correct Sciatic Nerve Management to Apply Ultrasound-Guided Percutaneous Neuromodulation in Patients With Chronic Low Back Pain: A Pilot Study. Neuromodulation. 2021 Aug;24(6):1067-1074. doi: 10.1111/ner.13396. Epub 2021 Apr 20. PMID 33876885
- [Background] Borrella-Andres S, Malo-Urries M, Perez-Bellmunt A, Arias-Buria JL, Rodriguez-Sanz J, Albarova-Corral MI, Gonzalez-Rueda V, Gallego-Sendarrubias GM, Fernandez-de-Las-Penas C, Lopez-de-Celis C. Application of Percutaneous Needle Electrolysis Does Not Elicit Temperature Changes: An In Vitro Cadaveric Study. Int J Environ Res Public Health. 2022 Nov 26;19(23):15738. doi: 10.3390/ijerph192315738. PMID 36497812
- [Background] Calderon-Diez L, Sanchez-Sanchez JL, Robles-Garcia M, Belon-Perez P, Fernandez-de-Las-Penas C. Cadaveric and Ultrasound Validation of Percutaneous Electrolysis Approach at the Achilles Tendon as a Potential Treatment for Achilles Tendinopathy: A Pilot Study. Int J Environ Res Public Health. 2022 Sep 21;19(19):11906. doi: 10.3390/ijerph191911906. PMID 36231206
- [Background] Munoz-Fernandez AC, Barragan-Carballar C, Villafane JH, Martin-Perez S, Alonso-Perez JL, Diaz-Meco R, Garcia-Jimenez D, Sanchez-Romero EA. A new ultrasound-guided percutaneous electrolysis and exercise treatment in patellar tendinopathy: three case reports. Front Biosci (Landmark Ed). 2021 Nov 30;26(11):1166-1175. doi: 10.52586/5017. PMID 34856761